CLINICAL TRIAL: NCT00101036
Title: A Phase II Study of GW572016 (Lapatanib) in Locally Advanced or Metastatic Hepato-Biliary Cancers
Brief Title: Lapatinib in Treating Patients With Locally Advanced or Metastatic Biliary Tract or Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03065; NCI-2012-03065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-53 (Other: UC Davis Comprehensive Cancer Center); 6674 (Other: CTEP); N01CM62201 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well lapatinib works in treating patients with locally advanced or metastatic biliary tract or liver cancer that cannot be removed by surgery. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The goal of this study is to determine the objective response rate of GW572016 in patients with biliary cancer and hepatocellular cancer (HCC).

SECONDARY OBJECTIVES:

I. Determine the overall survival of patients entered onto study. II. Quantitative and qualitative toxicities of the patient population treated with GW572016.

III. Determine the progression free survival of patients. IV. To perform molecular and pharmacogenomic correlative studies that will identify specific patient subsets that benefit from GW572016 therapy.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor site (biliary tree cancer [includes ampullary, bile duct, and gall bladder cancer] vs hepatocellular cancer).

Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed, surgically unresectable biliary cancer (gallbladder, ampullary, intra or extrahepatic bile duct) OR patients must have surgically unresectable HCC and who are not candidates for percutaneous ethanol injection or radio frequency ablation (RFA); patients must have histological or cytological confirmation of HCC
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan; if a patient has undergone TACE, ethanol or RFA ablation then new lesions need to be present in the liver, if there are no other sites of disease
* Patients may have received prior therapy as follows:

  * No more than one prior chemotherapy regimen for metastatic or recurrent disease will be allowed; prior chemotherapy for earlier stage disease (neoadjuvant, adjuvant, or concurrent with radiation therapy) will be allowed in addition to prior chemotherapy for recurrent metastatic disease; TACE is considered one regimen; at least 3 weeks must have elapsed since prior therapy, and toxicities of therapy should have resolved to =< Grade 1
  * Patients may have received prior radiation therapy; three weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all toxicities; measurable disease must either be outside the previous radiation field, or progressing within a radiated field, or a new lesion must be present
  * There must be no plans for the patient to receive concurrent hormonal, biologic, or radiation therapy to measurable lesions
  * Patients who have had prior treatment with EGFR targeting therapies are ineligible
  * Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy
* Life expectancy of greater than 12 weeks
* ECOG performance status less than or equal to 2 (Karnofsky >= 60%)
* Patients who have scores that fall into Childs B or C groups are excluded
* Patients must have organ and marrow function as defined below:
* Leukocytes >= 3000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Total bilirubin < 2 mg/dl
* AST(SGOT)/ALT(SGPT) =< 5.0 X upper limit of institutional normal (ULN)
* PT prolongation < 4 secs above ULN (unless taking warfarin)
* Creatinine =< ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Cardiac ejection fraction above the lower limit of normal as measured by echocardiogram or MUGA scan; note that baseline and on- treatment scans should be performed using the same modality and preferably at the same institution
* Adherence to the requirements for concomitant medications classified as CYP3A4 inducers or inhibitors
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with GW572016; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients requiring oral anticoagulants (coumadin, warfarin) are eligible provided there is appropriate close INR monitoring is in place; if medically appropriate and treatment available, the investigator may also consider switching these patients to low molecular weight (LMW) heparin, where an interaction with GW572016 is not expected
* The effects of GW572016 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Pregnant women are excluded from this study because GW572016 is member of the 4-anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GW572016, breastfeeding should be discontinued if the mother is treated with GW572016
* Ability to understand and the willingness to sign a written informed consent document
* Able to swallow and retain oral medication
* Patients with known brain metastases (Scans are not necessary to exclude brain metastasis) should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, will be excluded
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis) are also ineligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016 (i.e inhibitors of EGF and HER2- /neu) will render patients ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Ramanathan, Principal Investigator — UC Davis Comprehensive Cancer Center
Locations (1):
- UC Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: GW572016 1500 mg orally daily for 28 days, Biliary strata
- Arm 2: GW572016 1500 mg orally daily for 28 days, HCC strata
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 17 | 40
Completed | 17 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 17 | 40 | 57
Age, Continuous [Median (Full Range); unit: years] | 58 [44 to 76] | 62 [19 to 82] | 62 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 4 | 32 | 36
Region of Enrollment [Number; unit: participants]
  United States | 17 | 40 | 57

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT, MRI or X-Ray: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 5 years
Measure: Number; unit: percentage of responding patients
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 17 | 40
percentage of responding patients | 0 | 5

2. Secondary Outcome: Overall Survival
Description: Estimated by the Kaplan-Meier method.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 17 | 40
Months | 5.2 [3.3 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 6.2 [5.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Progression-free Survival
Description: Estimated using the Kaplan-Meier method. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 17 | 40
Months | 1.8 [1.7 to 5.2] | 2.3 [1.7 to 5.6]

4. Secondary Outcome: Disease Control Rate.
Description: The mathematical sum of percentages of complete response, partial response and stable disease.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 17 | 40
percentage of participants | 26 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 2 years, 3 months.
Description: "Other" adverse events include all grades and attribution to treatment that are not included in the "Serious" adverse events table.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 6/17 | 13/40
Other Adverse Events (participants affected / at risk) | 17/17 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=17) | Arm 2 (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 4 (4)
Fever (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (3)
Bone infection (Infections and infestations) | 1 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperbilirubinemia (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=17) | Arm 2 (N=40)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (9) | 20 (67)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (9)
Abdominal pain (Gastrointestinal disorders) | 4 (8) | 15 (25)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (5) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 10 (12) | 26 (58)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 6 (17)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 4 (7)
Nausea (Gastrointestinal disorders) | 9 (23) | 20 (32)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (8) | 9 (11)
Chest pain (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 14 (14) | 22 (22)
Edema limbs (General disorders) | 0 (0) | 5 (8)
Fatigue (General disorders) | 12 (21) | 27 (68)
Fever (General disorders) | 2 (2) | 2 (3)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
General symptom (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 2 (2)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 4 (6) | 18 (46)
Alkaline phosphatase increased (Investigations) | 9 (15) | 18 (44)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (8) | 26 (91)
Creatinine increased (Investigations) | 1 (1) | 5 (8)
Hyperbilirubinemia (Investigations) | 7 (9) | 15 (40)
INR increased (Investigations) | 1 (2) | 4 (6)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Leukopenia (Investigations) | 0 (0) | 5 (18)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Lymphopenia (Investigations) | 2 (4) | 7 (13)
Neutrophil count decreased (Investigations) | 0 (0) | 5 (7)
Platelet count decreased (Investigations) | 0 (0) | 12 (42)
Weight loss (Investigations) | 3 (4) | 7 (8)
Anorexia (Metabolism and nutrition disorders) | 5 (11) | 16 (23)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (17) | 20 (50)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8) | 15 (31)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 4 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5) | 3 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6) | 12 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 5 (6)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (3)
Taste alteration (Nervous system disorders) | 2 (3) | 6 (9)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Confusion (Psychiatric disorders) | 1 (2) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 7 (10)
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (10)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (5) | 9 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (10)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 10 (16)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (5) | 12 (37)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (17)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less